CLINICAL TRIAL: NCT01439633
Title: Pilot Study to Evaluate OFDI Surveillance and Image Guided Biopsy of the Esophagus
Brief Title: Optical Frequency Domain Imaging (OFDI) Surveillance and Image Guided Biopsy of the Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-P-000553; 2R01CA103769-06A1 (NIH)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Esophagus; OCT; Imaging
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGH OFDI marking and imaging (Experimental): OFDI imaging
  Interventions: Device: MGH OFDI marking

INTERVENTIONS:
Device: MGH OFDI marking — Imaging of esophagus with OFDI system

SUMMARY:
The specific aim of this study is to determine the feasibility of marking target pathologic locations identified on Optical Frequency Domain Imaging (OFDI) datasets using superficial cautery marks of the esophagus that are visible by endoscopy for subsequent guidance of biopsy.

DETAILED DESCRIPTION:
Twenty four consenting patients undergoing esophagogastroduodenoscopy (EGD) surveillance following a confirmed diagnosis of Barrett's esophagus will be recruited at Massachusetts General Hospital (MGH) . Along with Optical Frequency Domain Imaging (OFDI) imaging and cautery marking for targeted biopsy, the patients will undergo a standard of care clinical Esophagogastroduodenoscopy (EGD) procedure including endoscopic random biopsy. This study requires the use of a balloon catheter which is a commonly used technique and is accepted in clinical practice for dilation of esophageal and colonic strictures and for photodynamic therapy.

Once in position, the OFDI tissue marking laser will be activated by the physician. The physician will control the marking and make two marks of a duration of 2 seconds each. The 2 seconds time period will limit the tissue effects to only the superficial layers of the esophageal mucosa.

It is expected that the total experimental time including insertion and inflation of the OFDI balloon catheter, OFDI imaging, tissue marking, and removal of the OFDI balloon will add approximately 15 minutes to the total length of the EGD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an EGD for Barrett's esophagus surveillance with a prior confirmed Barrett's segment at least 1 cm in length
* Patients must be over the age of 18
* Patient must be able to give informed consent
* Women with child bearing potential must have a negative pregnancy test prior to procedure

Exclusion Criteria:

* Patients on anti-platelet and anti-coagulation medications and NSAIDS at the time of procedure
* Patients with a history of hemostasis disorders
* Patients that are pregnant
* Patients with esophageal strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD PhD, Principal Investigator — Massachusetts General Hospital; Norman Nishioka, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Suter MJ, Gora MJ, Lauwers GY, Arnason T, Sauk J, Gallagher KA, Kava L, Tan KM, Soomro AR, Gallagher TP, Gardecki JA, Bouma BE, Rosenberg M, Nishioka NS, Tearney GJ. Esophageal-guided biopsy with volumetric laser endomicroscopy and laser cautery marking: a pilot clinical study. Gastrointest Endosc. 2014 Jun;79(6):886-96. doi: 10.1016/j.gie.2013.11.016. Epub 2014 Jan 23. PMID 24462171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGH OFDI Marking and Imaging
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty two subjects were enrolled and twenty two finished completed this study
Arm/Group | MGH OFDI Marking and Imaging
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in Which the Targeted Locations Identified Through OFDI Imaging Correlates With the Biopsies.
Description: Determination of the feasibility to mark targeted pathologic locations identified through OFDI imaging using superficial cautery marks.Verification by endoscopy and utilization of the marks for biopsy guidance.Images will be analyzed and compared to biopsies of the correlated marked tissue.
Time Frame: day 1, during diagnostic procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MGH OFDI Marking and Imaging
Number analyzed (Participants) | 22
Participants | 22

ADVERSE EVENTS:
Arm/Group | MGH OFDI Marking and Imaging
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No